CLINICAL TRIAL: NCT06963294
Title: The Effect of Intraoperative Ketamine and Dexmedetomidine Use on Postoperative Delirium and Cognitive Dysfunction in Patients Undergoing Total Joint Arthroplasty
Brief Title: Ketamine and Dexmedetomidine for Delirium in Joint Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. prof, Haseki Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Haseki berna
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Delirium; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Saline Infusion (Placebo Comparator): Participants receive 0.9% saline at 30 mL/hour during surgery.
  Interventions: Drug: Ketamine
- Ketamine Infusion (Experimental): Participants receive ketamine at 0.1 mg/kg/hour as intraoperative infusion
  Interventions: Drug: Ketamine
- Dexmedetomidine Infusion (Experimental): Participants receive dexmedetomidine at 0.5 mcg/kg/hour as intraoperative infusion
  Interventions: Drug: Ketamine
- Ketamine + Dexmedetomidine (Experimental): Participants receive a combination of ketamine (0.3 mg/kg/hour) and dexmedetomidine (0.5 mcg/kg/hour) as intraoperative infusion.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Ketamine will be administered as an intravenous infusion at 0.1 mg/kg/hour during surgery

SUMMARY:
This prospective, randomized, double-blind, placebo-controlled clinical trial aims to evaluate the effects of intraoperative ketamine and dexmedetomidine on the incidence of postoperative delirium (POD) and postoperative cognitive dysfunction (POCD) in patients undergoing total joint arthroplasty. Given the high incidence of neurocognitive complications in elderly patients following major orthopedic surgeries, neuroprotective strategies during anesthesia are of growing interest. Both ketamine and dexmedetomidine have shown potential in reducing neuroinflammation and improving postoperative cognitive outcomes in previous studies.

Eighty adult patients (ASA I-III, aged 18-100) scheduled for elective total hip or knee arthroplasty under spinal anesthesia will be randomized into four groups: control (saline infusion), ketamine infusion, dexmedetomidine infusion, and combined ketamine + dexmedetomidine. Cognitive assessments will be performed preoperatively and on postoperative days 2 and 15 using the Mini Mental State Examination (MMSE). Delirium assessments will be conducted using the Confusion Assessment Method (CAM) postoperatively on days 1, 3, and 15.

Secondary outcomes include perioperative levels of cortisol, CRP, and fibrinogen, as well as postoperative pain scores (VAS) and analgesic consumption. The results are expected to clarify whether intraoperative administration of ketamine or dexmedetomidine can reduce the incidence of POD/POCD and improve postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective total joint arthroplasty (hip or knee)
* ASA physical status I-III
* Age between 18 and 100 years
* Ability to provide informed consent and comply with cognitive assessments

Exclusion Criteria:

* Pre-existing cognitive dysfunction or diagnosed neurodegenerative disease
* Hearing or language impairment interfering with MMSE/CAM evaluation
* Known allergy to ketamine or dexmedetomidine
* Significant cardiac arrhythmia (e.g., supraventricular tachycardia, 2nd or 3rd degree AV block)
* Renal insufficiency (GFR <30 mL/min/1.73 m²)
* Severe hepatic dysfunction

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-05-05 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Cognitive Dysfunction (POCD) Measured by MMSE | Baseline (preoperative), Postoperative Day 2, and Postoperative Day 15
  Cognitive function will be assessed using the Mini Mental State Examination (MMSE). A decrease of ≥2 points from baseline will be considered indicative of POCD.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hovaguimian F, Tschopp C, Beck-Schimmer B, Puhan M. Intraoperative ketamine administration to prevent delirium or postoperative cognitive dysfunction: A systematic review and meta-analysis. Acta Anaesthesiol Scand. 2018 Oct;62(9):1182-1193. doi: 10.1111/aas.13168. Epub 2018 Jun 26. PMID 29947091
- [Result] Singh A, Brenna CTA, Broad J, Kaustov L, Choi S. The Effects of Dexmedetomidine on Perioperative Neurocognitive Outcomes After Cardiac Surgery: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Ann Surg. 2022 May 1;275(5):864-871. doi: 10.1097/SLA.0000000000005196. Epub 2021 Aug 27. PMID 35543164